CLINICAL TRIAL: NCT00005766
Title: Clinical Trial of Creatine in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00109-0750; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Creatinine

INTERVENTIONS:
Drug: Creatinine

SUMMARY:
The objective of this study is to determine whether creatine slows disease progression in subjects with amyotrophic lateral sclerosis (ALS). ALS is a progressive uniformly lethal neurodegenerative disorder for which there is no known cure. Recent genetic and biochemical studies implicate free radical toxicity, glutamate excitotoxicity and mitochondrial dysfunction as possible causes of familial ALS (FALS) and sporadic ALS (SALS). It has been hypothesized that in ALS there may be involvement of oxidative free radical damage and impaired mitochondrial energy metabolism that could in turn lead to excitotoxic cell death. Creatine, an agent that improves mitochondrial function, has been shown to be neuroprotective in animal models of ALS and Huntington's disease.

This study is a double-blind, randomized, placebo-controlled trial of the safety and efficacy of creatine in patients with ALS enrolled at sites distributed throughout the United States, including Northeast ALS (NEALS) sites. The study will provide preliminary data on the safety and efficacy of creatine in ALS. If creatine slows disease progression in ALS and is well tolerated, a phase 3 study with survival as the primary outcome measure will be initiated.

114 eligible subjects will be randomized to receive treatment for 6 months of (1) active creatine or (2) placebo. After randomization, subjects will be followed prospectively for 6 months. The primary outcome measure for the study is the change in upper extremity motor function after 6 months of experimental therapy as tested with the Tufts Quantitative Neuromuscular Exam. Strength in eight arm muscles will be measured (bilateral shoulder and elbow flexion and extension). Secondary outcome measures include grip strength, motor unit number estimates (MUNE), the ALS functional rating score-revised (ALSFRS-R), and rate of change of a well established biochemical marker of oxidative damage to DNA (8OH2'dG levels in urine), and the safety and tolerability of creatine.

ELIGIBILITY:
Inclusion Criteria:

* ALS
* FVC >=50%
* Abnormality in upper and/or lower extremity motor function
* Not pregnant
* Disease duration <5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States